CLINICAL TRIAL: NCT06804174
Title: Distinct Endometrial Protein Profiles in Spontaneous and Stimulated Cycles in Women With Poor Ovarian Respons
Brief Title: Comparison of Endometrial Protein Profile in Spontaneous Versus Stimulated Menstrual Cycles in Poor Responders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (ARRS) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: (0120-319/2021/3)
Record Dates: First submitted 2025-01-27; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-10

CONDITIONS: Proteome
Keywords: endometrium, proteome, poor ovarian response, spontaneous cycle, stimulated cycle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Poor responder women as per POSEIDON criteria (Experimental)
  Interventions: Other: use of gonadotropins

INTERVENTIONS:
Other: use of gonadotropins — Comparison of endometrial proteome during the window of implantation between stimulated and spontaneous cycles.

SUMMARY:
Evaluation of endometrial protein profile in spontaneous and stimulated menstrual cycles

ELIGIBILITY:
Inclusion Criteria:

1. Primary infertility
2. Poor ovarian response

Exclusion Criteria:

1. Normal or high ovarian response to gonadotropin stimulation
2. Menstrual cycle disorders
3. Severe male cause of infertility
4. Preimplantation genetic testing
5. Pathological findings of the uterus (fibroids, endometrial polyps, adenomyosis) and fallopian tubes (distal occlusion of one or both fallopian tubes with hydrosalpinx).

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with poor ovarian response
Enrollment: 15 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Analysis of endometrial proteome after the use of gonadotropins | From enrollment to the end of treatment (approximately 2 months).
  Comparison of endometrial proteome during the window of implantation between spontaneous and stimulated cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Prof. Vrtačnik bokal, MD, PhD, Study Chair — Division of Obstetrics and Gynecology, University Medical Centre Ljubljana
Locations (1):
- Division of Obstetrics and Gynecology, university Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided